CLINICAL TRIAL: NCT00481247
Title: An Open-Label, Randomized, Multicenter Phase III Trial of Dasatinib (SPRYCEL®) vs. Standard Dose Imatinib (400 mg) in the Treatment of Subjects With Newly Diagnosed Chronic Phase Philadelphia Chromosome Positive Chronic Myeloid Leukemia
Brief Title: A Phase III Study of Dasatinib vs Imatinib in Patients With Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia
Acronym: DASISION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-056; 2006-005712-27 (EudraCT Number)
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: Chronic Phase Philadelphia Chromosome Positive Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasatinib (Experimental)
  Interventions: Drug: Dasatinib
- Imatinib (Active Comparator)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, oral, dasatinib 50-140 mg once daily (QD)
  Other Names: Sprycel®; BMS-354825
  Arms: Dasatinib
Drug: Imatinib — Tablets, oral, imatinib 200-800 mg, QD
  Arms: Imatinib

SUMMARY:
The purpose of this clinical research study is to compare the confirmed complete cytogenetic response of dasatinib with that of imatinib within 12 months after randomization in patients with newly diagnosed chronic-phase Philadelphia positive chronic myeloid leukemia. The safety of this treatment will also be studied.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, aged 18 years and older
* Chronic phase, Philadelphia Chromosome-positive chronic myeloid leukemia (CML)
* Eastern Cooperative Oncology Group Performance Status score of 0-2

Key Exclusion Criteria:

* Pleural Effusion
* Uncontrolled cardiovascular disease
* Significant bleeding disorder unrelated to CML
* Prior treatment with interferon/imatinib/dasatinib/anti-CML systemic treatments except anagrelide/hydroxyurea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (97):
- Molecular Md, Portland, Oregon, United States
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
- Australia (4):
  - Local Institution, Waratah, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Perth, Western Australia
- Austria (2):
  - Local Institution, Innsbruck
  - Local Institution, Vienna
- Belgium (2):
  - Local Institution, Bruges
  - Local Institution, Brussels
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, São Paulo, São Paulo
- Local Institution, Santiago, Santiago Metropolitan, Chile
- China (4):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Fuzhou, Fujian
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Tianjin, Tianjin Municipality
- Colombia (2):
  - Local Institution, Colombia, Bogota D.C.
  - Local Institution, Bogotá
- Czechia (4):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Olomouc
  - Local Institution, Prague
- Local Institution, Aarhus, Denmark
- France (12):
  - Local Institution, Nantes, Cedex 1
  - Local Institution, Brest
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Poitiers
  - Local Institution, Rennes
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Rostock
  - Local Institution, Tübingen
  - Local Institution, Ulm
- Local Institution, Thessaloniki, Greece
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Debrecen
- India (5):
  - Local Institution, Vellore, Tamil Nadu
  - Local Institution, Ahmedabad
  - Local Institution, Kochi
  - Local Institution, Mumbai
  - Local Institution, Trivandrum
- Italy (6):
  - Local Institution, Bologna
  - Local Institution, Catania
  - Local Institution, Monza (mb)
  - Local Institution, Orbassano (to)
  - Local Institution, Pavia
  - Local Institution, Roma
- Japan (12):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kamogawa-shi, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Morioka, Iwate
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Shinagawa-ku, Tokyo
- Mexico (4):
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Mexico, D. F., Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Culiacán, Sinaloa
- Netherlands (2):
  - Local Institution, Groningen
  - Local Institution, Nijmegen
- Peru (2):
  - Local Institution, Arequipa, Arequipa
  - Local Institution, Lima, Lima Province
- Poland (5):
  - Local Institution, Chorzów
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Rostov-on-Don
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- Local Institution, Seoul, South Korea
- Spain (7):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Oviedo
  - Local Institution, Salamanca
  - Local Institution, Valencia
- Turkey (Türkiye) (2):
  - Local Institution, Ankara
  - Local Institution, Kayseri

REFERENCES:
- [Derived] Glauche I, Kuhn M, Baldow C, Schulze P, Rothe T, Liebscher H, Roy A, Wang X, Roeder I. Quantitative prediction of long-term molecular response in TKI-treated CML - Lessons from an imatinib versus dasatinib comparison. Sci Rep. 2018 Aug 17;8(1):12330. doi: 10.1038/s41598-018-29923-4. PMID 30120281
- [Derived] Hughes TP, Saglio G, Quintas-Cardama A, Mauro MJ, Kim DW, Lipton JH, Bradley-Garelik MB, Ukropec J, Hochhaus A. BCR-ABL1 mutation development during first-line treatment with dasatinib or imatinib for chronic myeloid leukemia in chronic phase. Leukemia. 2015 Sep;29(9):1832-8. doi: 10.1038/leu.2015.168. Epub 2015 Jun 29. PMID 26118315
- [Derived] Fujisawa S, Nakamae H, Ogura M, Ishizawa K, Taniwaki M, Utsunomiya A, Matsue K, Takamatsu Y, Usuki K, Tanimoto M, Ishida Y, Akiyama H, Onishi S. Efficacy and safety of dasatinib versus imatinib in Japanese patients with newly diagnosed chronic-phase chronic myeloid leukemia (CML-CP): Subset analysis of the DASISION trial with 2-year follow-up. Int J Hematol. 2014 Feb;99(2):141-53. doi: 10.1007/s12185-013-1470-1. Epub 2013 Dec 20. PMID 24357015
- [Derived] Jabbour E, Kantarjian HM, Saglio G, Steegmann JL, Shah NP, Boque C, Chuah C, Pavlovsky C, Mayer J, Cortes J, Baccarani M, Kim DW, Bradley-Garelik MB, Mohamed H, Wildgust M, Hochhaus A. Early response with dasatinib or imatinib in chronic myeloid leukemia: 3-year follow-up from a randomized phase 3 trial (DASISION). Blood. 2014 Jan 23;123(4):494-500. doi: 10.1182/blood-2013-06-511592. Epub 2013 Dec 5. PMID 24311723
- [Derived] Kantarjian HM, Shah NP, Cortes JE, Baccarani M, Agarwal MB, Undurraga MS, Wang J, Ipina JJ, Kim DW, Ogura M, Pavlovsky C, Junghanss C, Milone JH, Nicolini FE, Robak T, Van Droogenbroeck J, Vellenga E, Bradley-Garelik MB, Zhu C, Hochhaus A. Dasatinib or imatinib in newly diagnosed chronic-phase chronic myeloid leukemia: 2-year follow-up from a randomized phase 3 trial (DASISION). Blood. 2012 Feb 2;119(5):1123-9. doi: 10.1182/blood-2011-08-376087. Epub 2011 Dec 9. PMID 22160483
- [Derived] Kantarjian H, Shah NP, Hochhaus A, Cortes J, Shah S, Ayala M, Moiraghi B, Shen Z, Mayer J, Pasquini R, Nakamae H, Huguet F, Boque C, Chuah C, Bleickardt E, Bradley-Garelik MB, Zhu C, Szatrowski T, Shapiro D, Baccarani M. Dasatinib versus imatinib in newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2010 Jun 17;362(24):2260-70. doi: 10.1056/NEJMoa1002315. Epub 2010 Jun 5. PMID 20525995
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 547 patients enrolled, 519 were randomized and 516 received treatment. Of the 28 who were enrolled but not randomized, 20 no longer met study criteria, 3 withdrew consent, 1 was lost to follow-up, and 4 withdrew for other reasons.
Groups:
- Dasatinib: Tablets, oral, dasatinib 100 mg once daily (QD)
- Imatinib: Tablets, oral, imatinib 400mg once daily (QD)
Period: Overall Study
Arm/Group | Dasatinib | Imatinib
Started | 259 (Randomized) | 260 (Randomized)
Received Treatment | 258 | 258
Completed | 0 | 0
Not Completed | 259 | 260
Not completed — Death | 0 | 1
Not completed — Disease progression | 18 | 22
Not completed — Intolerance | 42 | 17
Not completed — Treatment failure | 10 | 14
Not completed — AE unrelated to study drug | 13 | 4
Not completed — Withdrawal by Subject | 8 | 13
Not completed — Pregnancy | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Poor compliance/noncompliance | 1 | 7
Not completed — Administrative reason by sponsor | 157 | 162
Not completed — Varied | 6 | 15
Not completed — Did not receive treatment | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Imatinib: Tablets, oral, imatinib 400 mg once daily (QD)
- Total: Total of all reporting groups
Arm/Group | Dasatinib | Imatinib | Total
Number analyzed (Participants) | 259 | 260 | 519
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (14.6) | 47.1 (13.9) | 46.7 (14.2)
Age, Customized [Number; unit: Participants]
  <20 years | 5 | 9 | 14
  Between 21 and 45 years | 123 | 102 | 225
  Between 46 and 65 years | 111 | 125 | 236
  Between 66 and 75 years | 13 | 20 | 33
  >75 years | 7 | 4 | 11
Gender [Count of Participants; unit: Participants]
  Female | 115 | 97 | 212
  Male | 144 | 163 | 307
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 132 | 143 | 275
  Black/African American | 2 | 1 | 3
  Asian | 108 | 95 | 203
  Other | 17 | 21 | 38
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG is a 6-item scale used to assess disease progression, daily functioning, and appropriate treatment and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all predisease performance without restriction and (worst score) 5=death.
  Participants
    ECOG score=0 | 213 | 205 | 418
    ECOG score=1 | 46 | 53 | 99
    ECOG score=2 | 0 | 2 | 2
Number of Patients With Liver Involvement [Number; unit: Participants] | 37 | 18 | 55
Number of Participants With Spleen Involvement [Number; unit: Participants] | 83 | 71 | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Confirmed Complete Cytogenetic Response (cCCyR) Within 12 Months
Description: Cytogenetic response (CyR) is based on the prevalence of Philadelphia positive (Ph+) cells in metaphase from bone marrow (BM) sample. (Ideally, 25 metaphases but at least 20 metaphases from a BM sample were evaluated). Complete Cytogenetic Response (CCyR)=0% Ph+ cells in metaphase in BM. A cCCyR=those in which all measurements up to at least 28 days after the initial response show an equivalent or better CCyR.
Time Frame: Pretreatment, every 3 months up to 12 months
Population: All randomized participants
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 259 | 260
Participants | 204 | 177
Statistical Analysis 1: Comparison: Dasatinib vs Imatinib; Test type: Superiority or Other; p = 0.0056, Cochran-Mantel-Haenszel — A priori threshold for statistical significance=0.05; Cochran-Mantel-Haenszel test stratified by Hasford Score

2. Secondary Outcome: Percentage of Participants Remaining in Confirmed Complete Cytogenetic Response (cCCyR)
Description: Cytogenetic response (CyR) is based on the prevalence of Philadelphia positive (Ph+) cells in metaphase from bone marrow (BM) sample. (Ideally, 25 metaphases but at least 20 metaphases from a BM sample were evaluated). Complete Cytogenetic Response (CCyR)=0% Ph+ cells in metaphase in BM. A cCCyR=those in which all measurements up to at least 28 days after the initial response show an equivalent or better CCyR.
  Percentage of participants in cCCyR at years 2, 3, 4 and 5 was computed for all randomized participants who achieved cCCyR as measured from the time of first confirmation until the date of progression or death. Participants with cCCyR who neither progress nor die are censored on the date of their last cytogenetic assessment. Participants without cCCyR are considered to have progressed on Day 1.
Time Frame: Years 2, 3, 4 and 5
Population: All randomized participants who achieved cCCyR
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 215 | 204
percentage of participants
  At Year 2 | 98.0 [94.7 to 99.2] | 96.9 [93.2 to 98.6]
  At Year 3 | 96.9 [93.3 to 98.6] | 95.7 [91.6 to 97.8]
  At Year 4 | 95.6 [91.4 to 97.8] | 95.7 [91.6 to 97.8]
  At Year 5 | 93.1 [86.5 to 96.5] | 91.0 [83.6 to 95.2]
Statistical Analysis 1: Comparison: Dasatinib vs Imatinib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.55 to 1.13]

3. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Any Time
Description: Molecular response was assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction. MMR is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale (ie, at least 3 log reduction from a standardized baseline value).
Time Frame: Planned total follow-up duration of 5 years
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 259 | 260
Percentage of participants | 76.4 | 64.2

4. Secondary Outcome: Time to Confirmed Complete Cytogenic Response (cCCyR) Overall
Description: The time to cCCyR for all randomized participants is defined as the time from the randomization date until criteria are first met for complete cytogenic response (provided it is confirmed later). The time to cCCyR analysis censors nonresponders who do not progress at their last cytogenetic assessments and nonresponders who progress at the maximum time of all randomized participants.
  .
Time Frame: Day 1 to 5 years
Population: All randomized participants who achieved cCCyR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 215 | 204
Months | 3.1 [3.0 to 3.1] | 5.8 [5.6 to 6.0]
Statistical Analysis 1: Comparison: Dasatinib vs Imatinib; Hazard Ratio and Confidence Interval were based on analyses on all randomized subjects; Test type: Superiority or Other; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [1.20 to 1.77]

5. Secondary Outcome: Time to Major Molecular Response (MMR) Overall
Description: The time to MMR for all randomized participants is defined as the time from randomization date until measurement criteria are first met for MMR. The time to MMR analysis censors nonresponders who do not progress at their last molecular assessments and nonresponders who progress at the maximum time of all randomized participants.
Time Frame: Day 1 to 5 years
Population: All participants who received treatment and achieved MMR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 198 | 167
Months | 9.3 [8.8 to 11.8] | 15.0 [12.2 to 18.2]
Statistical Analysis 1: Comparison: Dasatinib vs Imatinib; Hazard Ratio, and Confidence Interval were based on analyses on all randomized subjects; Test type: Superiority or Other; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [1.25 to 1.89]

6. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization until progression (any progression/death within 30 days of last dosing date, or between 30-60 days of last dosing prior to start of secondary therapy). Those who did not progress/die or who progressed/died after 60 days of last dose were censored at last on-study hematologic/cytogenetic assessment; those with progression/death 30-60 days of last dosing date and after start date of secondary therapy censored at last on-study hematologic/cytogenetic assessment prior to start of secondary therapy; those who had not received study treatment censored on date randomized.
Time Frame: Participants were followed-up for at least 5 years
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 259 | 260
Percentage of participants | 88.9 | 89.2

7. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death. If the participant had not died, survival was censored on last date the participant was known to be alive.
Time Frame: Participants were followed-up for at least 5 years
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 259 | 260
Percentage of participants | 90.9 | 89.6

8. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs), Drug-related AEs, Drug-related Serious Adverse Events (SAEs), Drug-related AEs Leading to Discontinuation, and All Deaths
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From date of last person, first visit to date of last person, last visit (approximately 8 years)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 258 | 258
Participants
  All AEs | 251 | 251
  All Drug-related AEs | 224 | 231
  Diarrhea | 100 | 91
  Pleural effusion | 74 | 3
  Nausea | 40 | 74
  Cough | 68 | 28
  Muscle spasms | 14 | 63
  Thrombocytopenia | 61 | 50
  Neutropenia | 60 | 49
  Headache | 59 | 46
  Pyrexia | 58 | 51
  Vomiting | 43 | 54
  SAEs | 90 | 70
  Drug-related SAEs | 43 | 22
  AEs leading to discontinuation | 51 | 26
  All deaths | 26 | 26

9. Other Pre Specified Outcome: Number of Participants With Grade 3/4 Abnormalities in On-study Laboratory Test Results
Description: ULN=upper limit of normal. Grade 3=Severe AE; Grade 4=Life-threatening or disabling AE. Absolute neutrophil count: Grade 3 <1000-500/mm^3; Grade 4 <500/mm^3. Hemoglobin: Grade 3 <8.0-6.5 g/dL; Grade 4 <6.5 g/dL. Platelets: Grade 3 <50,000-25,000/mm^3; Grade 4 <25,000/mm^3. ALT/AST: Grade 3 >5.0-20*ULN; Grade 4 >20*ULN. Total bilirubin: Grade 3 >3-10*ULN; Grade 4 >10*ULN. Sample normal ranges (may vary by institution): ALT, Female: 7-30 U/L, Male: 10-55 U/L; AST, Female: 9-25 U/L, Male10-40 U/L; Total bilirubin: 0.0-1.0 mg/dL. Creatinine: Grade 3 >3.0-6.0*ULN; Grade 4 >6.0*ULN. Phosphate: Grade 3 <2.0-1.0 mg/dL; Grade 4 <1.0 mg/dL. Calcium: Grade 3 <7.0-6.0 mg/dL; Grade 4 <6.0 mg/dL. Potassium: Grade 3 <3.0-2.5 mmol/L; Grade 4 <2.5 mmol/L.
Time Frame: From date of last person, first visit to date of last person, last visit (approximately 8 years)
Population: Participants with laboratory assessments
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 256 | 257
Participants
  Grade 3/4 Absolute neutrophil count | 74 | 61
  Grade 3/4 Hemoglobin | 35 | 23
  Grade 3/4 Platelets | 56 | 37
  Grade 3/4 Alanine aminotransferase (ALT) | 2 | 4
  Grade 3/4 Aspartate aminotransferase (AST) | 2 | 3
  Grade 3/4 Total bilirubin | 3 | 0
  Grade 3/4 Creatinine | 3 | 2
  Grade 3/4 Phosphate | 19 | 79
  Grade 3/4 Calcium | 9 | 7
  Grade 3/4 Potassium | 0 | 8

ADVERSE EVENTS:
Time Frame: Randomization to end of study (December 2015)
Description: Study initiated: September 2007; End of Study: December 2015
Arm/Group | Dasatinib | Imatinib
Serious Adverse Events (participants affected / at risk) | 90/258 | 70/258
Other Adverse Events (participants affected / at risk) | 216/258 | 231/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=258) | Imatinib (N=258)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 1
BICYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1
SINOATRIAL BLOCK (Cardiac disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
HYPERTENSIVE CARDIOMEGALY (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
PERICARDITIS (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0
GLAUCOMA (Eye disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 0 | 1
SCLERAL HAEMORRHAGE (Eye disorders) | 1 | 0
CATARACT (Eye disorders) | 0 | 2
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 1
COLITIS (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 5 | 3
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
ILEUS (Gastrointestinal disorders) | 2 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0
PROTEIN-LOSING GASTROENTEROPATHY (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 3
FATIGUE (General disorders) | 2 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
OEDEMA (General disorders) | 0 | 1
PYREXIA (General disorders) | 3 | 2
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
CHRONIC GASTRITIS (Gastrointestinal disorders) | 1 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PANCREATIC DISORDER (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
DEVICE OCCLUSION (General disorders) | 1 | 0
PAIN (General disorders) | 1 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 0
ABSCESS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 0
CELLULITIS (Infections and infestations) | 3 | 0
ERYSIPELAS (Infections and infestations) | 2 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 1
INFECTION (Infections and infestations) | 3 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2
MENINGOENCEPHALITIS BACTERIAL (Infections and infestations) | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 3 | 3
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 2 | 2
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 0 | 1
H1N1 INFLUENZA (Infections and infestations) | 1 | 0
HEPATITIS VIRAL (Infections and infestations) | 0 | 1
MENINGITIS VIRAL (Infections and infestations) | 1 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
SKIN INJURY (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 0 | 1
KLEBSIELLA TEST POSITIVE (Investigations) | 1 | 0
TRANSAMINASE INCREASED (Investigations) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
JAW CYST (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
BLAST CELL PROLIFERATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
OPTIC NEURITIS (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLAST CELL IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NODAL MARGINAL ZONE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 13 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 7 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 1 | 0
URINARY BLADDER POLYP (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
UROGENITAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
SCROTAL OEDEMA (Reproductive system and breast disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1
HAEMORRHAGE (Vascular disorders) | 0 | 1
PHLEBITIS (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCULUSIVE DISEASE (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=258) | Imatinib (N=258)
ANAEMIA (Blood and lymphatic system disorders) | 38 | 31
LEUKOPENIA (Blood and lymphatic system disorders) | 21 | 28
NEUTROPENIA (Blood and lymphatic system disorders) | 60 | 49
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 59 | 48
EYELID OEDEMA (Eye disorders) | 7 | 40
PERIORBITAL OEDEMA (Eye disorders) | 4 | 20
ABDOMINAL PAIN (Gastrointestinal disorders) | 36 | 28
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 22 | 18
CONSTIPATION (Gastrointestinal disorders) | 21 | 7
DIARRHOEA (Gastrointestinal disorders) | 99 | 89
DYSPEPSIA (Gastrointestinal disorders) | 17 | 22
GASTRITIS (Gastrointestinal disorders) | 23 | 18
NAUSEA (Gastrointestinal disorders) | 40 | 74
VOMITING (Gastrointestinal disorders) | 41 | 52
ASTHENIA (General disorders) | 42 | 37
CHEST PAIN (General disorders) | 24 | 13
FACE OEDEMA (General disorders) | 14 | 27
FATIGUE (General disorders) | 40 | 40
INFLUENZA LIKE ILLNESS (General disorders) | 17 | 13
OEDEMA (General disorders) | 10 | 24
OEDEMA PERIPHERAL (General disorders) | 25 | 32
PYREXIA (General disorders) | 58 | 50
TOOTHACHE (Gastrointestinal disorders) | 17 | 10
INFLUENZA LIKE ILLNESS (General disorders) | 23 | 17
NASOPHARYNGITIS (Infections and infestations) | 32 | 43
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 30 | 28
HAEMOGLOBIN DECREASED (Investigations) | 30 | 17
WEIGHT INCREASED (Investigations) | 25 | 33
BRONCHITIS (Infections and infestations) | 20 | 14
CONJUNCTIVITIS (Infections and infestations) | 10 | 17
GASTROENTERITIS (Infections and infestations) | 19 | 10
INFLUENZA (Infections and infestations) | 20 | 12
URINARY TRACT INFECTION (Infections and infestations) | 11 | 13
ALANINE AMINOTRANSFERASE INCREASE (Investigations) | 13 | 7
DECREASED APPETITE (Metabolism and nutrition disorders) | 23 | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 34 | 38
BACK PAIN (Musculoskeletal and connective tissue disorders) | 34 | 44
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 14 | 63
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 22 | 19
MYALGIA (Musculoskeletal and connective tissue disorders) | 36 | 39
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 28 | 39
DIZZINESS (Nervous system disorders) | 28 | 18
HEADACHE (Nervous system disorders) | 59 | 46
INSOMNIA (Psychiatric disorders) | 20 | 16
DEPRESSION (Psychiatric disorders) | 5 | 13
COUGH (Respiratory, thoracic and mediastinal disorders) | 68 | 28
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 36 | 10
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 69 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 15 | 19
RASH (Skin and subcutaneous tissue disorders) | 45 | 44
ACNE (Skin and subcutaneous tissue disorders) | 14 | 1
PALLOR (Vascular disorders) | 7 | 13
HYPERTENSION (Vascular disorders) | 26 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.